CLINICAL TRIAL: NCT06025227
Title: Provide Pre-approval Single Patient Expanded Access (Compassionate Use) of Etrasimod for Patients.
Status: Available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C504
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Etrasimod — tablets

SUMMARY:
Provide pre-approval single patient Expanded Access (Compassionate Use) of Etrasimod for patients.

DETAILED DESCRIPTION:
In Expanded Access, treating physicians are the Sponsors. Expanded Access requests from treating physicians may be submitted to www.pfizercares.com. Availability will depend on location and country.

ELIGIBILITY:
Patient must be intolerant, have a contraindication or had inadequate response to at least 3 therapies available for Ulcerative Colitis (UC) in this country or provide a rationale of why therapy was not used.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult